CLINICAL TRIAL: NCT03080480
Title: Efficacy and Safety of Pioglitazone Therapy for Chronic Granulomatous Disease Patients With Severe Infection.
Brief Title: Pioglitazone Therapy for Chronic Granulomatous Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The results are negtive.
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinqiao Sun, Professor, Children's Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTSICGD
Record Dates: First submitted 2017-02-27; First posted 2017-03-15 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic Granulomatous Disease; Severe Infection; PPARγ; Pioglitazone; phagocytes
MeSH Terms: conditions — Granulomatous Disease, Chronic; Infections | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pioglitazone (Experimental): Treatment for chronic granulomatous disease patients with severe infection.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone is PPARγ agonist that may be enhance ROS production and partially restore host phagocytes in CGD.
  pioglitazone is administered at a starting dose of 1 mg/kg and given the absence of adverse effects is progressively increased up to 3 mg/kg or 30 mg/daily.
  Other Names: ACTOS

SUMMARY:
The purpose of this proposed research is to investigate the efficacy and safety of the therapy with pioglitazone for chronic granulomatous disease (CGD) patients severe infection.

DETAILED DESCRIPTION:
Chronic granulomatous disease (CGD) is a rare genetic disease caused by defects in genes encoding the subunits of the nicotinamide adenine dinucleotide（NADPH）phosphate oxidase complex. In normal phagocytes peroxisome proliferator-activated receptor gamma (PPARγ) activation links NADPH oxidase activity with enhanced mitochondrial reactive oxygen species (ROS) production. There is deficient mitochondrial ROS production in CGD，due to the lack of this upstream signaling by the NADPH oxidase and PPARγ. These patients are susceptible to bacterial and fungal infections, as well as extensive tissue granuloma formation. X-chromosome-linked CGD (X-CGD) is most frequently. And it generally produces a severe phenotype, with a mortality rate of 3% to 5% per year despite state-of-the-art prophylaxis and intensive multimodal treatment.

At present the most curative treatment for patients with X-CGD is hematopoietic stem cell transplantion (HSCT). But for many patients without an HLA-matched donor and active infections/inflammatory complications still require novel approches.

PPARγ agonist such as pioglitazone, approved for type 2 diabetes, was reported to bypass the need for the NADPH oxidase for enhanced mtROS production and partially restored host defense in CGD. What's more, some animal models and several clinical cases have proved its efficacy. The investigators propose to study the efficacy and safety of the therapy with pioglitazone for children with severe infection of CGD, and its long-term effects.

Through this study the investigators hope to confirm the benefits of pioglitazone in the treatment of this rare disease especially for those patients without a prompt suitable matched donor or for whom the critical disease conditions force to postpone HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age：1 months to 18 years
2. Chronic Granulomatous Disease
3. with severe infections

Exclusion Criteria:

1. > 18 years of age
2. infections are treatable by conventional therapy (antibiotics, antimycotics, allogeneic granulocytes)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
efficiency of Pioglitazone | 3 years
  Frequency of infections as indicator for the drug's benefit for the patients; Functional reconstitution of the NADPH oxidase in circulating cells of the peripheral blood (Stimulation Index by DHR analysis).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 3 years
  Frequency and severity of metabolic disorders and unexpected toxic adverse events during and after using pioglitazone

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Migliavacca M, Assanelli A, Ferrua F, Cicalese MP, Biffi A, Frittoli M, Silvani P, Chidini G, Calderini E, Mandelli A, Camporesi A, Milani R, Farinelli G, Nicoletti R, Ciceri F, Aiuti A, Bernardo ME. Pioglitazone as a novel therapeutic approach in chronic granulomatous disease. J Allergy Clin Immunol. 2016 Jun;137(6):1913-1915.e2. doi: 10.1016/j.jaci.2016.01.033. Epub 2016 Apr 4. No abstract available. PMID 27056268
- [Background] Fernandez-Boyanapalli RF, Falcone EL, Zerbe CS, Marciano BE, Frasch SC, Henson PM, Holland SM, Bratton DL. Impaired efferocytosis in human chronic granulomatous disease is reversed by pioglitazone treatment. J Allergy Clin Immunol. 2015 Nov;136(5):1399-1401.e3. doi: 10.1016/j.jaci.2015.07.034. Epub 2015 Sep 18. No abstract available. PMID 26386811
- [Background] Fernandez-Boyanapalli RF, Frasch SC, Thomas SM, Malcolm KC, Nicks M, Harbeck RJ, Jakubzick CV, Nemenoff R, Henson PM, Holland SM, Bratton DL. Pioglitazone restores phagocyte mitochondrial oxidants and bactericidal capacity in chronic granulomatous disease. J Allergy Clin Immunol. 2015 Feb;135(2):517-527.e12. doi: 10.1016/j.jaci.2014.10.034. Epub 2014 Dec 10. PMID 25498313
- [Derived] Hui X, Liu D, Wang W, Hou J, Ying W, Zhou Q, Yao H, Sun J, Wang X. Low-Dose Pioglitazone does not Increase ROS Production in Chronic Granulomatous Disease Patients with Severe Infection. J Clin Immunol. 2020 Jan;40(1):131-137. doi: 10.1007/s10875-019-00719-z. Epub 2019 Nov 19. PMID 31745699